CLINICAL TRIAL: NCT03289000
Title: A Retrospective Study to Evaluate the ConforMIS iTotal® Posterior Stabilized (PS) Knee Replacement System
Status: Completed | Type: Observational
Sponsor: Restor3D (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-004
Record Dates: First submitted 2017-09-15; First posted 2017-09-20 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Osteo Arthritis Knee
Keywords: osteoarthritis; knee arthroplasty; knee replacement; patient specific
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- ConforMIS PS Group: Patients who have undergone a total knee replacement with the ConforMIS iTotal PS Knee Replacement System
  Interventions: Device: iTotal Posterior Stabilized (PS) Knee Replacement System

INTERVENTIONS:
Device: iTotal Posterior Stabilized (PS) Knee Replacement System — Patient-specific posterior stabilized total knee replacement and patient specific surgical jigs

SUMMARY:
This study is a retrospective, multi-center study, with one single remote follow up contact. This study will include a minimum of 80 patients and a maximum 100 patients who have been treated with the ConforMIS iTotal PS knee product.

DETAILED DESCRIPTION:
Patients will be contacted either by phone or email for a single remote follow-up. Retrospective data will be collected from medical records including pre-operative, operative and any follow up visits which have occurred since implantation as available. . All data will be collected from existing medical records and from single follow up call/email.

* Demographics and Medical History
* Pre & Post-Operative Data including Range of Motion
* Surgical Data
* Survivorship (phone/email or last known visit)
* Patient Reported Outcomes (phone/email single time point visit)

  * Patient Satisfaction
  * KOOS Jr.

ELIGIBILITY:
Inclusion Criteria:

1. Previously underwent surgical implantation of a ConforMIS iTotal PS knee replacement.
2. Over 18 Years of age

Exclusion Criteria:

1. BMI > 40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who are 18 years or older and have received a ConforMIS iTotal PS knee replacement to treat any condition indicated on the device's instructions for use.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2017-08-04 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Demographics and Medical History | 1 year
  Demographics and medical history gathered from medical records
Pre and Post Operative Range of Motion | 1 year
  Collected retrospectively through medical records, collecting range of motion from pre-operative visits and post-operative visits

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Tennessee Orthopaedic Alliance, Nashville, Tennessee
  - Scott Orthopedic Center, Huntington, West Virginia